CLINICAL TRIAL: NCT02246244
Title: Randomized, Double Blind, Efficacy Study of Escitalopram Versus Placebo in ENT Cancer Patients Suffering From Emotional Distress
Brief Title: Randomized, Double Blind, Efficacy Study of Escitalopram in ENT Cancer Patients Suffering From Emotional Distress
Acronym: TADDOR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2008-002159-25; 2008/1388 (Other: CSET number)
Record Dates: First submitted 2014-09-17; First posted 2014-09-22 (Estimated); Last update posted 2016-06-10 (Estimated); Status verified 2016-06

CONDITIONS: ENT Cancer
MeSH Terms: interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Escitalopram (Experimental): 10 mg once per day
  Interventions: Drug: Escitalopram
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Escitalopram
  Arms: Escitalopram
Other: Placebo
  Arms: Placebo

SUMMARY:
Escitalopram is an antidepressant inhibitor of the serotonin reuptake. On the market in France since 2002.

Prevalence of emotional distress in patients with cancer is 30-50%. this prevalence may vary regarding the tumor localisation, the population, intensity of the symptoms...

Incidence of ENT cancer is highly significant in France, it is one of the most important in the world 37 out of 100 000. it is in patients with ENT cancer that the prevalence of depression is the most important (22%-57%).

Researches appears necessary to assessed the efficacy of antidepressant treatments with as primary objective not only the decrease of depressive symptoms but also an ensemble of physic and psychological symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ENT cancer of stage I to IVb that have to go under surgery and/or radiotherapy and/or chemotherapy as first line treatment. It may be a primary cancer or a new localisation.
* Total score on HADS scale >11
* Patients aged from 18 to 75 years
* Signed informed consent
* OMS < 2, hospitalized or ambulatory
* Are authorized to inclusion, psychoactive treatments at stable dosage for two weeks for benzodiazepins, neuroleptics, antihistaminics or other anxiolytics or hypnotics

Exclusion Criteria:

* Patients in palliative treatments
* Previous bipolar disorder or schizophrenia
* Major depressive episode with severity criteria
* Suicidal patients
* Acute infection
* ASAT/ALAT >3N
* Creatinine clearance <30 ml/mn
* Natremia inferior to the laboratory standard
* For alcoholic patients non abstinent at the time of inclusion, previous "delirium tremens"
* Previous upper gist bleeding
* Inefficacy or intolerance of previous treatment by escitalopram
* Not compatible concomitant treatment:
* Other antidepressive than escitalopram (except clonazepam)
* all hypnotics (except zolpidem)
* all anxiolytics (except clonazepam, clorazepate and diazepam)
* medical treatment for smoking addiction like bupropion or varenicline
* Pregnant or breastfeeding women
* Patients under guardianship
* Patients without insurance
* Impossibility to follow the protocol for geographical, social or psychic reasons
* Insufficient knowledge of French

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2009-04; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Efficacy of treatment by Escitalopram on depressive symptoms | Assessed 3 months after randomization
  Assessed using HADS scale

SECONDARY OUTCOMES:
Efficacy of treatment on emotional distress | Assessed 3 months after randomization
  Assessed using HADS scale

CONTACTS AND LOCATIONS:
Locations (1):
- Gustave Roussy, Villejuif, Val de Marne, France

REFERENCES:
- [Derived] Vita G, Compri B, Matcham F, Barbui C, Ostuzzi G. Antidepressants for the treatment of depression in people with cancer. Cochrane Database Syst Rev. 2023 Mar 31;3(3):CD011006. doi: 10.1002/14651858.CD011006.pub4. PMID 36999619